CLINICAL TRIAL: NCT05177198
Title: Clinical and Radiographic Effects of Modified Minimally Invasive Surgical Technique With Clindamycin Augmented Platelet-rich Fibrin Versus Platelet-rich Fibrin Alone for Management of Periodontal Intrabony Defects: A Randomized Controlled Clinical Trial
Brief Title: Effects of Modified Minimally Invasive Surgical Technique With Clindamycin Augmented Platelet-rich Fibrin Versus Platelet-rich Fibrin Alone for Management of Periodontal Intrabony Defects.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Yusri El-Sayed El-Ashry, Masters Student at Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER332
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2021-12

CONDITIONS: Periodontal Intrabony Defects
Keywords: modified minimally invasive; Clindamycin; platelet-rich fibrin; intrabony defects
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (M-MIST + Clindamycin augmented PRF) (Experimental): Patients will be selected with probing pocket depth PD ≥ 5 mm and clinical attachment level (CAL) ≥ 5 mm, with vertical defects as detected in periapical radiographs will be treated with modified minimally invasive surgical technique with Clindamycin (at concentration of 150 mg/ml) augmented platelet-rich fibrin.
  Interventions: Procedure: M-MIST + Clindamycin augmented PRF
- Control group (M-MIST + PRF) (Experimental): Patients will be selected with probing pocket depth PD ≥ 5 mm and clinical attachment level (CAL) ≥ 5 mm, with vertical defects as detected in periapical radiographs will be treated with modified minimally invasive surgical technique with platelet-rich fibrin alone .
  Interventions: Procedure: M-MIST + PRF

INTERVENTIONS:
Procedure: M-MIST + Clindamycin augmented PRF — modified minimally invasive surgical technique with Clindamycin (at concentration of 150 mg/ml) augmented platelet-rich fibrin.
  Arms: Test group (M-MIST + Clindamycin augmented PRF)
Procedure: M-MIST + PRF — modified minimally invasive surgical technique with platelet-rich fibrin alone.
  Arms: Control group (M-MIST + PRF)

SUMMARY:
Periodontal infections in the oral cavity are strongly associated with clinical outcomes of both regenerative and conventional surgical procedures and should receive proper attention. It is evident with the available data that PRF has antimicrobial activity against microbial pathogens. Clindamycin is an effective antibiotic against anaerobic bacteria and it achieves higher levels of antimicrobial activity than other antibiotics. The use of PRF alone or in combination with other biomaterials (such as pharmacologic agents) provided safe and promising results in the form of improvements in clinical and radiographic parameters in the management of periodontal osseous defects.

DETAILED DESCRIPTION:
Many factors had to be taken into consideration while treating intrabony defects to achieve the concept of periodontal regeneration. PRF is a material that contains growth factors enmeshed in the fibrin network resulting in their sustained release over a period of time that can accelerate the wound healing process. The use of PRF alone or in combination with other biomaterials (such as pharmacologic agents) provided safe and promising results in the form of improvements in clinical and radiographic parameters in the management of periodontal osseous defects. The purpose of combination between the PRF and Clindamycin is for establishing a simple and practical method that gives antimicrobial properties to PRF and to provide evidence of its effectiveness, and that this may provide additional advantage and reduces the need for systemic antibiotics in a variety of oral surgical procedures. Protection of the regenerating area should be provided through the specifically designed surgical approaches. These different surgical approaches developed over time include differences in terms of flap design and suturing technique. Therefore, successful wound healing was strongly influenced by preservation of the microvasculature of soft tissues as well as by revascularization rates. The Minimally Invasive Surgical Technique (MIST) was proposed by to draw the aspects of wound and blood clot stability and primary wound closure for blood-clot protection. These concepts were further strengthened with the Modified Minimally Invasive Surgical Technique M-MIST, that further incorporated the concept of space provision for the process of regeneration. For this, the effect of Clindamycin augmented PRF together with M-MIST on the clinical and radiographic outcomes in the treatment of periodontal intrabony defects need to be evaluated for clinical effectiveness

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria:

  * Patient consulting in the outpatient clinic.
  * Able to tolerate surgical periodontal procedures.
  * Patient ready to perform oral hygiene instructions.
  * Compliance with the maintenance program.
  * Provide informed consent.
  * Accepts the 12 months follow-up period.
* Teeth related criteria:

  * Mature permanent tooth.
  * Tooth with two or three-walled intra-bony defect, with CAL ≥ 5mm and intra osseous defect ≥ 3mm.

Exclusion Criteria:

* Patient-related criteria:

  * Medically compromised patients.
  * Pregnant or nursing women.
  * Uncooperative patients.
  * Smokers.
* Teeth related criteria:

  * Teeth with one wall intra-bony defect.
  * Teeth with supra-bony defects.
  * Teeth with grade II or III mobility.
  * Teeth with proximal carious defects or proximal faulty restorations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level ( CAL) | 9 months
  Measured from the CEJ to the bottom of the gingival sulcus.

SECONDARY OUTCOMES:
Probing Depth (PD) | 9 months
  Measured from the gingival margin to the bottom of the gingival sulcus.
Radiographic linear defect depth | 9 months
  Measured as the depth of intra-osseous defect from the alveolar crest to the defect base
Radiographic defect bone density | 9 months
  The region of interest (ROI) is outlined, through drawing an outline corresponding to the demarcating walls of the intra-osseous defect and mean grey values are calculated
Gingival recession | 9 months
  Measured from the CEJ to the most apical extension of the gingival margin.
Plaque index | 9 months
  Scores 0,1,2,3
Gingival index | 9 months
  Scores 0,1,2,3

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Yusri, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided